CLINICAL TRIAL: NCT06732310
Title: The Unique and Combined Effects of Prenatal and Early Childhood Programming on Child Maltreatment: Examining Mechanisms of Change
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 22-05-7238; R01HD114597 (NIH)
Record Dates: First submitted 2024-12-04; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Child Abuse; Intimate Partner Violence; Secondary Prevention; Parenting
Keywords: child abuse; child maltreatment; intimate partner violence; domestic violence; secondary prevention; parenting
MeSH Terms: interventions — exopolysaccharide, Pseudomonas

STUDY DESIGN:
Intervention Model Description: In pregnancy: Women who receive the PMEP complete a structured set of sessions delivered over the course of 5 weeks, each session lasts 2 hours in duration: (1) becoming a group & safety planning, (2) identifying and understanding sources of stress, (3) strategies to build resilience and resolve conflict, (4) perinatal health and infant care, and (5) positive parenting. Women who are not randomized to PMEP participate in a contact-equivalent, non-directive social support group.
  In early childhood: Each of the 5 RET sessions are 1 hour in duration. The program is manualized and each session includes teaching/review of skills, instructions/activity with rationale, reminiscing practice, and immediate video feedback by a family coach. Families who are not randomized to the RET condition will be mailed a kit containing 5 packets to be opened weekly. Each packet includes a family activity and a newsletter with parenting materials.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PMEP + ECM (Experimental): In pregnancy: PMEP
  In early childhood: enhanced case management
  Interventions: Behavioral: Pregnant Moms' Empowerment Program; Behavioral: Enhanced Case Management
- Pregnancy - Active Control + RET (Experimental): In pregnancy: Women who are not randomized to PMEP participate in a contact-equivalent, non-directive social support group.
  In early-childhood: Women participant in the RET.
  Interventions: Behavioral: Reminiscing and Emotion Training; Behavioral: Pregnancy - Active Control
- PMEP + RET (Experimental): In pregnancy: PMEP
  In early childhood: Reminiscing and Emotion Training Program
  Interventions: Behavioral: Pregnant Moms' Empowerment Program; Behavioral: Reminiscing and Emotion Training
- Pregnancy - Active Control + ECM (Active Comparator): In pregnancy: Women not randomized to PMEP will participate in a contact-equivalent, nondirective social support group.
  In early childhood: Families who are not randomized to the RET condition will be mailed a kit containing 5 packets to be opened weekly. Each packet includes a family activity and a newsletter with parenting materials.
  Interventions: Behavioral: Pregnancy - Active Control; Behavioral: Enhanced Case Management

INTERVENTIONS:
Behavioral: Pregnant Moms' Empowerment Program — Women who receive the PMEP complete a structured set of sessions delivered over the course of 5 weeks, each session lasts 2 hours in duration: (1) becoming a group & safety planning, (2) identifying and understanding sources of stress, (3) strategies to build resilience and resolve conflict, (4) perinatal health and infant care, and (5) positive parenting.
  Other Names: PMEP
  Arms: PMEP + ECM; PMEP + RET
Behavioral: Reminiscing and Emotion Training — Each of the 5 RET sessions are 1 hour in duration. The program is manualized and each session includes teaching/review of skills, instructions/activity with rationale, reminiscing practice, and immediate video feedback by a family coach.
  Arms: PMEP + RET; Pregnancy - Active Control + RET
Behavioral: Pregnancy - Active Control — Women who are not randomized to the PMEP participate in a contact-equivalent, nondirective social support group.
  Other Names: AC
  Arms: Pregnancy - Active Control + ECM; Pregnancy - Active Control + RET
Behavioral: Enhanced Case Management — Families randomized to this attentional control condition will receive enhanced case management. They will be mailed a kit containing 5 packets to be opened weekly. Each packet includes a family activity and a newsletter with parenting materials (e.g., Adventures in Parenting curriculum developed by NICHD) that were selected to not overlap with RET content (e.g., reading together, fitness, etc.). Using mothers' responses regarding access to resources on the Family Resource Scale (Dunst & Leet, 1987), which is completed during the baseline visit, mothers will also receive referrals to community resources for items rated as inadequate.
  Other Names: ECM
  Arms: PMEP + ECM; Pregnancy - Active Control + ECM

SUMMARY:
Child maltreatment and child exposure to adult intimate partner violence (IPV) often co-occur and are detrimental to the mental and physical health of children, yet few prevention programs address these intersecting forms of adversity using dual-generation approaches. The proposed study is a rigorous randomized controlled trial that uses a 2x2 factorial design to evaluate the potential synergistic benefits of delivering programming prenatally and during early childhood in order to support the mother-child relationship and ultimately prevent child maltreatment. If effective in preventing child maltreatment, these programs have the potential for high public health impact given that they are both cost-effective and readily scalable.

DETAILED DESCRIPTION:
The study will occur at two sites - the University of Notre Dame and the University of Memphis. A total of N=300 mother-child dyads will participate, with an equal number of dyads drawn from each site - Memphis, TN (n=115) and South Bend, IN (n=115). The sample will be composed of n=230 women and children drawn from an ongoing randomized clinical trial (RCT) of the PMEP (R01HD098092); during Year 1 of the current study, we will implement the PMEP RCT protocol with an additional n=70 women, for a total sample of N=300 families.

In order to be eligible for the PMEP trial arm, women must be: 18 years or older, pregnant (between 10 and 30 weeks), English speaking, and exposed to IPV in the past year. To be eligible for re-enrollment in the RET trial arm, women must have previously participated in the PMEP trial arm. Women who have a significant mental health disorder or cognitive impairment that precludes their ability to understand or participate in the intervention will be excluded. Mothers who have experienced miscarriage, infant death, or who no longer have custody of the child with whom they were pregnant with when they participated in the PMEP trial arm will be excluded from the intervention given that the RET trial arm requires active participation from both parent and child; if mothers, however, have had another child who was born after PMEP who is in the eligible age range, they may participate.

The primary objective of the current study is to evaluate the unique and combined effects of evidence-based prenatal (i.e., Pregnant Moms' Empowerment Program) and early childhood (i.e., Reminiscing and Emotion Training) programming to prevent child maltreatment.

Study hypotheses are tested in a 2x2 randomized controlled trial design, with four conditions: PMEP + early childhood control, PMEP + RET, prenatal control + RET, or prenatal and early childhood controls.

Enrollment will continue for approximately 3.5 years, with an expected enrollment rate of approximately 8 mother-child dyads per month. For mother-child dyads who participated in the RCT of the PMEP (n = 230) the expected duration of the RET arm will be approximately 11 months. For the mother-child dyads who will be newly enrolled into the PMEP trial arm as part of the proposed study, the expected duration of the PMEP arm is 16 months; when these children are 3-6 years old, they will participate in the RET arm for 11 months.

Women and children newly enrolled in the PMEP trial arm as part of the current study will complete eight assessments. These will include four PMEP trial arm assessments (baseline [T1], post-test [T2], 3 month post-partum follow-up [T3], and 12 month post-partum follow-up [T4]) and four more assessments (baseline [T5], post-test [T6], 3 month follow-up [T7], 6 month follow-up [T8]) completed as part of the RET trial arm. Dyads only participating in the RET trial arm will participate in the 4 RET assessments (i.e., T5-T8). Women will be compensated for each assessment and children will receive a small toy.

Primary outcome measures will include DCS records (gathered at T5, T8, and 12 month follow-up) coded using the Maltreatment Classification System, the Maternal Maltreatment Classification Interview, the Adult Adolescent Parenting inventory, the Child Abuse Potential Inventory, the Revised Conflict Tactics Scale, and Maternal Sensitivity (coded from observational data). A number of covariates will also be collected, including maternal mental health, childhood trauma and traumatic/major life events over the study period, child exposure to other forms of violence, child temperament, and social support.

For women randomized to receive the PMEP intervention, participation will include five group sessions that utilize interactive learning and group-based discussion to empower women to end intergenerational cycles of violence and develop skills for sensitive, responsive parenting. PMEP includes a structured set of sessions, each 2 hours in duration: (1) becoming a group and safety planning, (2) identifying and understanding sources of stress, (3) strategies to build resilience and resolve conflict, (4) perinatal health and infant care, and (5) positive parenting.

For women randomized to receive RET, participation in the program will include five virtual RET sessions that aim to promote a positive, nurturing parent-child relationship during early childhood through training in sensitive parent-child communication about children's emotions. RET sessions will be 1 hour in duration. The program is manualized and each session includes teaching/review of skills, instructions/activity with rationale, reminiscing practice, and immediate video feedback by a family coach.

ELIGIBILITY:
The sample will be composed of n=230 women and children drawn from an ongoing randomized clinical trial (RCT) of the PMEP (R01HD098092); during Year 1 of the current study, we will recruit an additional n=70 pregnant, IPV-exposed women and implement the PMEP RCT protocol with them, for a total sample of N=300 families.

In order to be eligible for the PMEP trial arm, women must be: 18 years or older, pregnant (between 10 and 30 weeks), English speaking, and exposed to IPV in the past year. To be eligible for re-enrollment in the RET trial arm, women must have previously participated in the PMEP trial arm. Women who have a significant mental health disorder or cognitive impairment that precludes their ability to understand or participate in the intervention will be excluded. Mothers who have experienced miscarriage, infant death, or who no longer have custody of the child with whom they were pregnant with when they participated in the PMEP trial arm will be excluded from the intervention given that the RET trial arm requires active participation from both parent and child; if, however, women have a child born after their participation in PMEP and who is in the study age range, they and their child may participate.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
DCS Records - Maltreatment Classification System | RET baseline (T5), 6 month follow-up (T8). 12 month follow-up
  DCS records will be coded using the Maltreatment Classification System (MCS; Barnett et al., 1993). The MCS utilizes operational criteria for determining the occurrence of subtypes of maltreatment. Subtype categories include sexual abuse, physical abuse, physical neglect, and emotional maltreatment.
Maternal Maltreatment Classification Interview | RET baseline (T5), 6 month follow-up (T8)
  MCS ratings will be supplemented by information obtained during the Maternal Maltreatment Classification Interview (MMCI; Cicchetti et al., 2002), a structured interview based on the MCS. It will be audiotaped and coded by two independent raters utilizing the same operational criteria as the MCS.
Maltreatment risk/Propensity | PMEP baseline [T1], PMEP immediate post-test [T2], PMEP 3 month post-partum follow-up [T3], PMEP 12 month post-partum follow-up [T4], RET baseline [T5], RET immediate post-test [T6], RET 3 month follow-up [T7], RET 6 month follow-up [T8]
  Mothers will complete the Child Abuse Potential Inventory (CAPI; Milner, 1986) and the Adult Adolescent Parenting Inventory (AAPI; Bavolek & Keene, 2001), both of which assess maltreatment propensity. A composite variable of maltreatment propensity/risk will be created by combining these indicators.
Intimate partner violence | PMEP baseline [T1], PMEP immediate post-test [T2], PMEP 3 month post-partum follow-up [T3], PMEP 12 month post-partum follow-up [T4], RET baseline [T5], RET immediate post-test [T6], RET 3 month follow-up [T7], RET 6 month follow-up [T8]
  others will complete the Revised Conflict Tactics Scale (CTS2) (Straus, Hamby, Boney-McCoy, & Sugarman, 1996; Straus, 1979), which assesses the severity of psychological, physical, and sexual violence in a dating, cohabiting, or marital relationship. This measure has the advantage of being able to be flexibly coded to gain information about IPV severity, frequency, and chronicity.
Maternal Sensitivity - perinatal period | PMEP 3 month post-partum follow-up [T3], PMEP 12 month post-partum follow-up [T4]
  Maternal sensitivity will be assessed in several observational contexts. At T3 and T4, mother-child dyads will participate in a 5-minute free play activity that will be coded using an established coding framework (Braungart-Rieker et al., 2014).
Maternal Sensitive Guidance - early childhood | RET baseline [T5], RET immediate post-test [T6], RET 3 month follow-up [T7], RET 6 month follow-up [T8]
  From T5-T8, maternal sensitive guidance will be assessed by following the Autobiographical Emotional Events Dialogue procedure (AEED; Koren-Kari e, Oppenheim, Haimovich, & Etzion-Carasso, 2003b).
Maternal Sensitivity - DPICS - early childhood | RET baseline [T5], RET immediate post-test [T6], RET 3 month follow-up [T7], RET 6 month follow-up [T8]
  Participants will also complete a 10-minute free play paradigm using an abbreviated Dyadic Parent-Child Interaction Coding System (DPICS; Eyeberg, et al., 2013). This free play will be coded for positive, neutral and negative patterns of parent-child communication.

SECONDARY OUTCOMES:
Positive Parenting Behavior | RET baseline (T5), RET immediate post-test (T6), 3 month follow-up (T7), 6 month follow-up (T8)
  Positive parenting behavior will be assessed using selected subscales of the Alabama Parenting Questionnaire - Preschool Version (Clerkin, et al., 2007).
Maternal emotional style | RET baseline (T5), RET immediate post-test (T6), 3 month follow-up (T7), 6 month follow-up (T8)
  Maternal emotion style will be assessed using the Maternal Emotional Style Questionnaire (Lagacé-Séguin' & Coplan' 2005).
Child Emotion Regulation | RET baseline (T5), RET immediate post-test (T6), 3 month follow-up (T7), 6 month follow-up (T8)
  Children's emotion regulation will be assess via parent report on the Emotion Regulation Checklist (Shields & Cicchetti, 1997).
Child Temperament - infancy | PMEP 12 month postpartum follow-up (T4)
  Child temperament will be collected as a covariate. Mothers will complete the Infant Behavior Questionnaire at T4 (Rothbart, et al., 2001) which assesses multiple aspects of early child temperament.
Child Temperament - early childhood | RET baseline (T5), RET immediate post-test (T6), RET 3 month follow-up (T7), RET 6 month follow-up (T8)
  Child temperament will be collected as a covariate. Mothers will complete the the Child Behavior Questionnaire at T5-T8 (Rothbart, et al., 2001) which assesses multiple aspects of early child temperament.
Child Adjustment | RET baseline (T5), RET immediate post-test (T6), RET 3 month follow-up (T7), RET 6 month follow-up (T8)
  Child adjustment will be assessed using the Child Behavior Checklist (Achenbach, 1999) at assessments T5-T8.

OTHER OUTCOMES:
Maternal Trauma History | PMEP baseline [T1], RET baseline [T5]
  Maternal exposure to lifetime trauma, including both interpersonal and non-interpersonal traumas, will be assessed using the Trauma History Questionnaire (Hooper et al., 2011) at baseline interviews [T1, T5].
Maternal Child Maltreatment History | RET baseline [T5]
  Women's history of child maltreatment, specifically, will be assessed using the Childhood Trauma Questionnaire (Berstein et al., 1997) at T5.
Maternal Social Support | PMEP baseline [T1], PMEP immediate post-test [T2], PMEP 3 month post-partum follow-up [T3], PMEP 12 month post-partum follow-up [T4], RET baseline [T5], RET immediate post-test [T6], RET 3 month follow-up [T7], RET 6 month follow-up [T8]
  Women's access to social supports (friends, family, neighborhood) will be assessed using the Lubben Social Network Scale (Lubben & Gironda, 2004). This scale been used with IPV-exposed women.
Mother Verbal Ability | RET immediate follow-up [T6; mother]
  RET is a verbally mediated intervention, so mother verbal ability will be included as a covariate in the analyses. Verbal ability will be assessed using the Peabody Picture Vocabulary Test - Fifth Edition (Dunn, 2018).
Maternal Mental Health - PTSD | PMEP baseline [T1], PMEP immediate post-test [T2], PMEP 3 month post-partum follow-up [T3], PMEP 12 month post-partum follow-up [T4], RET baseline [T5], RET immediate post-test [T6], RET 3 month follow-up [T7], RET 6 month follow-up [T8]
  Maternal PTSD will be assessed using the PTSD Checklist-Civilian 5 (Weathers, et al., 2013).
Maternal Mental Health - Depression | PMEP baseline [T1], PMEP immediate post-test [T2], PMEP 3 month post-partum follow-up [T3], PMEP 12 month post-partum follow-up [T4], RET baseline [T5], RET immediate post-test [T6], RET 3 month follow-up [T7], RET 6 month follow-up [T8]
  Maternal depression will be assessed using the Center for Epidemiological Studies Depression Scale (Radloff, 1977).
Child victimization | RET baseline (T5), RET immediate post-test (T6), RET 3 month follow-up (T7), RET 6 month follow-up (T8)
  This questionnaire is used in nationally representative surveillance studies (NatSCEV) and is a recommended tool for monitoring purposes relative to children's experiences of violence, in conjunction with formal, state-level data (Forston, et al., 2016). Children's exposure to other types of violence, outside of maltreatment (e.g., community violence) will be assessed using this tool.
Child Verbal Ability | RET baseline [T5] and RET 6 month follow-up [T8]
  RET is a verbally mediated intervention, so child verbal ability will be included as a covariate in the analyses. Verbal ability will be assessed using the Peabody Picture Vocabulary Test - Fifth Edition (Dunn, 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Miller-Graff, PhD, Principal Investigator — University of Notre Dame; Kathryn H Howell, PhD, Principal Investigator — University of Wisconsin, Madison; Kristin Valentino, PhD, Principal Investigator — University of Notre Dame
Locations (2):
- United States (2):
  - University of Notre Dame, Notre Dame, Indiana
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Participants were not consented for IPD sharing in the initial study. Study data are sensitive and some data is highly protected (e.g., DCS records).